CLINICAL TRIAL: NCT03725462
Title: Evaluation of Electrophysiological Signal Measured by Smart Textile CE-marked
Acronym: STREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017-A00648-45
Record Dates: First submitted 2018-10-12; First posted 2018-10-31 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardioskin (Experimental): Subjects performed a monitoring with Cardioskin. The performance is evaluated either by a comparison with a gold standard, either by a comparison with anterior version of Cardioskin, either by an opinion of an expert.
  Interventions: Device: Cardioskin
- Neuronaute (Experimental): Subjects performed a monitoring with Neuronaute. The performance is evaluated either by a comparison with a gold standard, either by a comparison with anterior version of Neuronaute, either by an opinion of an expert.
  Interventions: Device: Neuronaute

INTERVENTIONS:
Device: Cardioskin — Subjects have a monitoring with cardioskin and comparator
  Arms: Cardioskin
Device: Neuronaute — Subjects have a monitoring with Neuronaute and comparator
  Arms: Neuronaute

SUMMARY:
The aim is to evaluate the performance of Cardioskin and Neuronaute, two connected medical devices CE-marked, manufactured by Bioserenity.

It's an open monocentric comparative clinical study, where subjects will test the Cardioskin device and/or the Neuronaute device.

DETAILED DESCRIPTION:
With this study evulating the performance of two wireless, connected device of electrophysiological signal monitoring. The Cardioskin monitors electrocardiogram signal. The Neuronaute monitors electroencephalogram, electromyogram and electrocardiogram.

This study will permit to optimize the devices performance.

To the study, subjects of at least 18 years old will test Cardioskin and or Neuronaute device, without randomization.

ELIGIBILITY:
Inclusion Criteria:

• man or women of at least 18 years old

Exclusion Criteria:

* Injuries or wounds on the body and scalp
* Participant unable to follow the procedure of use, the judgment of the investigator
* Brain surgery that occurred less than a week ago
* Known allergy to silver, polyamide, silicone, synthetic materials
* Sensory disorders that make the subject insensitive to pain
* behavioral problems that make the subject excessively agitated or aggressive;
* Cardiorespiratory disorders that may be aggravated by mild compression of thorax
* Subject equipped with an electrical stimulation device;
* Inappropriate anthropometric parameters to textile sizes
* Clinically detectable or known pain of the subject;
* Current participation in a clinical trial or participation in a previous clinical study including a period of deficiency not yet completed at the time of this clinical trial
* Predisposition to tension headaches (the compression exerted by the cap may in some cases trigger a headache);
* Use of the Cardioskin device for resuscitation or intensive care.
* Participant with defibrillator, vagus nerve stimulator or other high frequency surgical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Sensor quality validation | 2 month
  Signal is considered as of "good quality" " not good quality" regarding criteria of signal patterns (eg.beat detection, beats variability..)

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, Paris, France